CLINICAL TRIAL: NCT00875173
Title: Selenium Treatment and Chagasic Cardiopathy (STCC): A Prospective Randomized Trial in Patients With Chagas Disease
Brief Title: Selenium Treatment and Chagasic Cardiopathy (STCC)
Acronym: STCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Tania Araujo-Jorge, Full Professor,MD, PhD, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oswaldo Cruz
Record Dates: First submitted 2008-10-20; First posted 2009-04-03 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Chagas Disease
Keywords: Selenium; Chagas disease; Chagasic cardiopathy
MeSH Terms: conditions — Chagas Disease | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selenium (Experimental): Sodium selenite 100 micrograms in capsugel by mouth diary for 365 consecutive days
  Interventions: Drug: Selenium
- Placebo (Active Comparator): Capsugel for placebo (selenium 100 micrograms capsugel) by mouth diary for 365 consecutive days
  Interventions: Drug: Placebo (for Selenium)

INTERVENTIONS:
Drug: Selenium — selenium as a drug according to Brazilian regulation laws
  Other Names: Antioxidant therapy
  Arms: Selenium
Drug: Placebo (for Selenium) — Placebo with similar flavor, smell and colour.
  Other Names: control
  Arms: Placebo

SUMMARY:
Background:

Chagasic myocardiopathy caused by the protozoa Trypanosoma cruzi has been the principal cause of cardiac death in Latin America. Without any trypanocidal therapeutic intervention, infected subjects can pass from the indeterminate to the cardiac form with heart dysfunction. Our group has studied the role and the effect of the supplementation with the essential micronutrient selenium (Se) on T. cruzi infection, and the investigators have verified that:

1. low Se levels is related to the severity of the myocardiopathy in chagasic patients
2. adequate Se diet is essential for mice survival at the acute phase of the experimental T. cruzi infection
3. Se supplementation prevented the myocardial lesions at the acute phase in mice. From these findings and considering that Se supplementation was able to prevent Keshan cardiopathy, to revert electrocardiographic and echocardiographic alterations in patients nourished by parenteral route, and reduced re-infarction and cardiac deaths from acute myocardial infarction; the investigators purpose to investigate if Se treatment via oral route, is able to impair the progress of heart dysfunction in chagasic patients expressed by the study of progression rate and by the comparison of the means of ventricular ejection fraction.

Methods:

The Selenium treatment and Chagasic Cardiopathy (STCC) trial is double-blind, placebo controlled, randomized in 130 chagasic patients at the chronic phase following the inclusion criteria of (a) altered ECHO (LVEF between 0,35 % and 45 %), (b) age between 20 and 65 years, (c) randomly divided in two groups: Placebo (n=65) and Se (n=65). Patients of Se group will intake diary 100 µg Se as sodium selenite for 12 months. The primary endpoint is the reduction of 50 % in the progression rate of heart dysfunction, and the secondary endpoint is a partial or total reversion in electrocardiography alterations.

Conclusion:

This trial was recently approved by Brazilian Research Ethics Committee and will be conducted in accordance with the principles for human experimentation. If the investigators confirmed the benefit of Se treatment, a strategy of utilization a micronutrient in an adequate concentration as a treatment in diary diet can revolutionize the therapeutic for chagasic myocardiopathy.

DETAILED DESCRIPTION:
Several induced cardiomyopathy , Mycoplasma pneumonia-induced myocarditis, heart damage investigations have shown positive effects of Se on experimental models: cardiotoxicity induced by chemotherapics, ischemic cardiopathy, CVB3 and LP-BM5 (murine AIDS, retrovirus)-in reperfused heart, and in chagasic cardiopathy. In addition, beneficial effects of Se supplementation were reported in patients with myocardial infarct, Keshan disease, and cardiac dysfunction during HPN.

Our group has investigated the role and Se effect on infection by T. cruzi. By evaluating plasma Se levels in 170 chagasic patients, we discovered that the frequency of subjects with Se levels lower than normal was significantly higher in those with severe cardiopathy. Moreover, in this pioneering research, we found a positive correlation between Se levels and the LVEF, indicating that normal Se levels pave the way for efficient cardiac function. Later, we investigated if nutritional deficiency of this trace element interfered with the development of cardiopathy and the susceptibility to experimental T. cruzi infection. In that study, we found 100 % of mortality in Se deficient mice, while in the selenium adequate groups only 20% of the male and no female died even at 40 dpi. In addition, parasitemia levels of infected mice were not altered by Se deficiency, suggesting that the high susceptibility at the acute phase was not due to the parasite load. We later investigated if Se treatment could minimize the course of T. cruzi infection or the myocarditis in mice. We verified that the concentration of 4 ppm Se did not alter the resistance to infection but was able in preventing the increase of CK-MB levels in infected mice, indicating that Se helps to protect the heart from inflammatory damage driven by T. cruzi infection.

Currently, experimental and clinical trials concerning Se supplementation have been performed; however, to date, there is no trial regarding the use of this micronutrient as a treatment to protect cardiac function in chagasic patients with cardiopathy. The present clinical trial aims to study the effect of Se intervention on the progression rate of the cardiopathy in patients with mild or moderate HD (LVEF between 35 % and 45 %) in order to validate this new strategy of treatment. The HD will be expressed by the progression rate and by the comparison of means of the LVEF. In this context we will test the hypothesis that Se treatment is able to interfere with the progression of cardiac dysfunction in chronic chagasic patients. We expect the impediment of the progression of ventricular dysfunction in patients with mild HD, and the improvement of cardiac function in patients with moderate HD in the group of patients receiving Se therapy. This is the first clinical trial concerning this specific group of cardiac chagasic patients with mild or moderate HD.

ELIGIBILITY:
Inclusion Criteria:

* altered ECHO (LVEF between 0,35 % and 45 %)
* age between 20 and 65 years

Exclusion Criteria:

* patients > 65 years of age
* smoke habit, patients with non-chagasic cardiopathy, live close to mineral deposit, metals industries and place with radioactive exposition, vegetarian
* depressive psychological profile
* pregnant or in lactating period
* present or presented cancer or diabetes.
* patients will be excluded if they take anti-convulsive medicines (Clozapine, Valproic Acid)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2008-10; Primary Completion 2016-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Ejection fraction by echocardiography | Twice a year

SECONDARY OUTCOMES:
Electrocardiography | twice a year

CONTACTS AND LOCATIONS:
Overall Officials: Tania C Araujo-Jorge, MD/PhD, Principal Investigator — Instituto Oswaldo Cruz
Locations (1):
- Instituto Nacional de Infectologia/Instituto de Pesquisa Clínica Evandro Chagas, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Holanda MT, Mediano MFF, Hasslocher-Moreno AM, Gonzaga BMS, Carvalho ACC, Ferreira RR, Garzoni LR, Pereira-Silva FS, Pimentel LO, Mendes MO, Azevedo MJ, Britto C, Moreira OC, Fernandes AG, Santos CM, Constermani J, Paravidino VB, Maciel ER, Carneiro FM, Xavier SS, Sperandio da Silva GM, Santos PF, Veloso HH, Brasil PEAA, de Sousa AS, Bonecini-de-Almeida MG, da Silva PS, Sangenis LHC, Saraiva RM, Araujo-Jorge TC. Effects of Selenium treatment on cardiac function in Chagas heart disease: Results from the STCC randomized Trial. EClinicalMedicine. 2021 Aug 28;40:101105. doi: 10.1016/j.eclinm.2021.101105. eCollection 2021 Oct. PMID 34485877
- [Derived] Holanda MT, Mediano MFF, Hasslocher-Moreno AM, Xavier SS, Saraiva RM, Sousa AS, Maciel ER, Carneiro FM, da Silva PS, Sangenis LHC, Veloso HH, Cardoso CSA, Bonecini-Almeida MDG, Souza AL, Roma EH, Azevedo MJ, Pereira-Silva FS, Pimentel LO, Mendes MO, Garzoni LR, Gonzaga BMS, Carvalho ACC, Brasil PEAA, Sperandio da Silva GM, Araujo-Jorge TC. A protocol update for the Selenium Treatment and Chagasic Cardiomyopathy (STCC) trial. Trials. 2018 Sep 19;19(1):507. doi: 10.1186/s13063-018-2889-8. PMID 30231899
- [Derived] Alvarenga Americano do Brasil PE, Pereira de Souza A, Hasslocher-Moreno AM, Xavier SS, Lambert Passos SR, de Fatima Ramos Moreira M, Santini de Oliveira M, Sperandio da Silva GM, Magalhaes Saraiva R, Santos de Aguiar Cardoso C, de Sousa AS, Mediano MF, Bonecini de Almeida Mda G, da Cruz Moreira O, Britto C, de Araujo-Jorge TC. Selenium Treatment and Chagasic Cardiopathy (STCC): study protocol for a double-blind randomized controlled trial. Trials. 2014 Oct 6;15:388. doi: 10.1186/1745-6215-15-388. PMID 25284194
- See also: Instituto Oswaldo Cruz — http://www.ioc.fiocruz.br